CLINICAL TRIAL: NCT06488573
Title: The Effect of a Nutritional Intervention Focused on Dietary Pattern in the Cardiovascular Risks of Individuals with Bipolar Disorder
Brief Title: PROgram to Enhance Cardiovascular Risk Trough an Intervention of Nutrition in Bipolar Disorder
Acronym: PROTECTION-BD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Deakin University (Other)
Responsible Party: Principal Investigator, Beny Lafer, Associated professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25299
Record Dates: First submitted 2024-06-17; First posted 2024-07-05 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Bipolar Depression; Bipolar Disorder (BD)
Keywords: nutrition intervention; nutritional psychiatry; bipolar disorder; dietary intervention; brazilian dietary guideline
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Intervention Model Description: Control group vs intervention group
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment as usual (No Intervention): Treatment as usual
- Nutritional intervention (Experimental): Nutritional intervention based on the Brazilian Dietary Guidelines
  Interventions: Behavioral: Nutritional intervention

INTERVENTIONS:
Behavioral: Nutritional intervention — 7 individual sessions + 8 small group sessions
  Arms: Nutritional intervention

SUMMARY:
Individuals with Bipolar Disorder (BD) have twice the risk of being affected by metabolic comorbidities and a 1.8-fold increased risk of mortality from cardiovascular diseases when compared to the general population. These factors are fundamental in the 14-year reduction in the life expectancy of people with TB reported in recent meta-analyses. This occurs mainly due to the increased inflammation associated with the disease, the adverse effects of pharmacological treatments and unhealthy lifestyle habits that are more common in people diagnosed with BD. Nutrition has been studied as an adjunctive treatment in other psychiatric disorders, but there is a lack of studies about the role of nutrition in TB. Considering that diet can impact metabolic health, this randomized controlled study aims to evaluate the effect of a nutritional intervention on cardiovascular risk in patients with TB. The intervention is based on the dietary pattern recommended in the Dietary Guidelines for the Brazilian Population and will be applied by a registered dietitian. According to the literature, the sample size will be 72 individuals with TB (36 in the control group with usual treatment + 36 in the intervention group added to the usual treatment). The intervention will be carried out in 7 individual sessions and 8 group sessions with specific themes. The primary aim of this protocol will be an intervention to contribute to cardiovascular health - verified by serum markers, anthropometric measurements and the Framingham Cardiovascular Risk Score (algorithm used to estimate an individual's 10-year cardiovascular risk). The secondary stages will be the adherence of the intervention and the impact on the quality of life of the participants. The possible positive results of this nutritional intervention can open new clinical perspectives. Meaning that might show that better food choices can protect the cardiovascular health of individuals with TB, leading to a reduction in morbidity and mortality associated with the disease.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Bipolar disorder types I and II diagnosis
* Adults of both genders, from 18 to 60 years old
* In typical pharmacotherapy for BD, for at least one month
* Agreement to participate in the study with signature of the consent form

Exclusion Criteria:

* Patients with "very good or excellent" diet quality assessed by the diet quality scale (ESQUADA): >275 out of a score of 375
* Patients in a state of hypomania or mania: score >8 (Young Mania Rating Scale - YMRS)
* Patients with severe depression >21 Montgomery-Åsberg Depression Rating Scale
* Patients at low cardiovascular risk (<7 points for men or <9 points for women on the Framingham Global Risk Score)
* Low weight or eutrophic body mass index: <25kg/m² as in similar studies
* Pregnant or breastfeeding women
* Patients diagnosed with anorexia and bulimia nervosa
* Patientes diagnosed with Irritable Bowl Syndrome or other diagnosed conditions that affect the gastrointestinal function

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
C reactive protein | Baseline, week 12, week 24 and follow up at week 52
  C reactive protein
Total cholesterol and fractions | Baseline, week 12, week 24 and follow up at week 52
  Total cholesterol and fractions
Glycemia | Baseline, week 12, week 24 and follow up at week 52
  Glycemia
Glycated hemoglobin A1C | Baseline, week 12, week 24 and follow up at week 52
  Glycated hemoglobin A1C
Triglycerides | Baseline, week 12, week 24 and follow up at week 52
  Triglycerides
HOMA IR | Baseline, week 12, week 24 and follow up at week 52
  HOME IR
Apoliporpotein B | Baseline, week 12, week 24 and follow up at week 52
  Apoliporpotein B
Cardiovascular risk | Baseline, week 12, week 24 and follow up at week 52
  Framingham Global Risk Score (-3 to 21; higher scores mean worse outcome)
Body weight | Baseline, week 12, week 24 and follow up at week 52
  Body weight
Body fat percentage | Baseline, week 12, week 24 and follow up at week 52
  Body fat percentage
waist circumference | Baseline, week 12, week 24 and follow up at week 52
  waist circumference

SECONDARY OUTCOMES:
Dietary assessment - dietary intake | Baseline, week 12, week 24 and follow up at week 52
  3-day food record from last week (calories and macronutrients)
Dietary assessment - dietary quality | Baseline, week 12, week 24 and follow up at week 52
  ESQUADA (0-375; higher scores mean better outcome)
Dietary assessment - dietary adehrence | Baseline, week 12, week 24 and follow up at week 52
  NUTRINET (0-72; higher scores mean worse outcome)
Quality of life WHOQOL | Baseline, week 12, week 24 and follow up at week 52
  WHOQOL Bref Portuguese (0-100; higher scores mean better outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Fernanda Gabriel, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided